CLINICAL TRIAL: NCT02608450
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Vehicle-Controlled Study to Evaluate the Safety and Efficacy of Cortexolone 17α-Propionate (CB-03-01) Cream, 1% Applied Twice Daily for 12 Weeks in Subjects With Facial Acne Vulgaris
Brief Title: A Study to Evaluate the Safety and Efficacy of CB-03-01 Cream, 1% in Subjects With Facial Acne Vulgaris (25)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cassiopea SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CB-03-01/25
Record Dates: First submitted 2015-11-17; First posted 2015-11-18 (Estimated); Results first posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Acne Vulgaris
Keywords: acne; clascoterone; anti-androgen
MeSH Terms: conditions — Acne Vulgaris | interventions — Clascoterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CB-03-01 cream (Experimental): CB-03-01 cream, 1% applied twice daily for 12 weeks
  Interventions: Drug: CB-03-01 cream, 1%
- Vehicle cream (Placebo Comparator): Vehicle cream applied twice daily for 12 weeks
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: CB-03-01 cream, 1% — CB-03-01 (cortexolone 17α-propionate) is a steroidal antiandrogen that is being developed as a 1% cream for the topical treatment of acne vulgaris.
  Other Names: cortexolone 17α-propionate; clascoterone (USAN, INN)
  Arms: CB-03-01 cream
Drug: Vehicle cream — Vehicle cream manufactured to mimic look and feel of CB-03-01 but without the active ingredient cortexolone 17α-propionate.
  Arms: Vehicle cream

SUMMARY:
The primary objective of this study is to determine the safety and efficacy of CB-03-01 cream, 1%, versus the vehicle cream applied twice daily for 12 weeks in subjects with facial acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or non-pregnant female, 9 years of age or older. Females must be post-menopausal, surgically sterile, or using highly effective birth control methods. Women of child-bearing potential must have a negative urine pregnancy test (UPT) at the Screening/Baseline Visit.
2. Subject has provided written and verbal informed consent/assent. A subject under 18 years of age must provide written informed assent and be accompanied by the parent or legal guardian at the time of assent/consent signing.
3. Subject has an Investigator's Global Assessment (IGA) score of 3 (moderate) or 4 (severe) [0 (clear) to 4 (severe) scale].
4. Subject has facial acne vulgaris with at least 30 to a maximum of 75 inflammatory lesions (papules, pustules, and nodules) and 30 to a maximum of 100 non-inflammatory lesions (open and closed comedones).
5. Subject and parent/guardian (if applicable) are willing to comply with study instructions and return to the clinic for required visits.
6. Subject has used the same type and brand of make-up, other facial products (exclusive of RX/OTC acne cleansers) and hair products (e.g., shampoo, gel, hair spray, mousse, etc.) for at least one (1) month prior to the Baseline Visit and agrees to continue his/her other general skin and hair care products and regimen for the entire study.

Exclusion Criteria:

1. Subject is pregnant, lactating, or is planning to become pregnant during the study.
2. Subject has any skin pathology or condition that could interfere with the evaluation of the test products or requires the use of interfering topical or systemic therapy.
3. Subject has greater than two (2) facial nodules.
4. Subject has nodulocystic acne.
5. Subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
6. Subject is currently enrolled in an investigational drug or device study.
7. Subject has received an investigational drug or has been treated with an investigational device within 30 days prior to the initiation of treatment (Baseline).
8. Subject has facial hair that could interfere with the study assessments in the opinion of the investigator.
9. Subject and parent/guardian (if applicable) are unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.
10. Subject may be unreliable for the study including subjects who engage in excessive alcohol intake or drug abuse, or subjects who are unable to return for scheduled follow-up visits.
11. Subject has known hypersensitivity or previous allergic reaction to any of the active or inactive components of the test articles.
12. Subject has the need or plans to be exposed to artificial tanning devices or excessive sunlight during the trial.
13. Subject has used any of the prohibited topical anti-acne treatments or procedures prior to the study unless appropriate washout period is documented.
14. Subject has used used any of the prohibited systemic anti-acne medications prior to the study unless appropriate washout period is documented.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 708 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R&D Cassiopea, Study Director — Cassiopea S.p.A.
Locations (54):
- United States (44):
  - Gary M. Petrus, MD PA, Little Rock, Arkansas
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - Vitiligo & Pigmentation Institute of Southern California, Los Angeles, California
  - San Diego Sports Medicine and Family Health Center, San Diego, California
  - Rady Childrens Hospital, Pediatric and Adolescent Dermatology, San Diego, California
  - Southern California Dermatology, Santa Ana, California
  - Clinical Science Institute, Santa Monica, California
  - Memorial Research Medical Clinic dba / Orange County Research Center, Tustin, California
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - Site 0190, Boca Raton, Florida
  - Study Protocol, Inc., Boynton Beach, Florida
  - Site 0196, Miami, Florida
  - Site 0197, Miami, Florida
  - Site 0198, Miami, Florida
  - Site 0199, Miami, Florida
  - Site 0191, Miami, Florida
  - Site 0192, Miami, Florida
  - Site 0195, Miami, Florida
  - Tory Sullivan, M.D., P.A., North Miami Beach, Florida
  - Meridien Research, St. Petersburg, Florida
  - MOORE Clinical Research, Inc., Tampa, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Site 0152, Carmel, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Henry Ford Health System, Detroit, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - The Center for Dermatology, Cosmetic & Laser Surgery, Mount Kisco, New York
  - DermResearch Center of New York, Inc., Stony Brook, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Oregon Dermatology and Research Center, Portland, Oregon
  - The Pennsylvania State University and the Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Greenville Dermatology, LLC, Greenville, South Carolina
  - International Clinical Research - Tennessee LLC, Murfreesboro, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Westlake Dermatology Clinical Research Center, Austin, Texas
  - Bellaire Dermatology Associates, Bellaire, Texas
  - J&S Studies, Inc., College Station, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - Clinical Research Associates of Tidewater, Inc., Norfolk, Virginia
  - Dermatology Associates, Seattle, Washington
  - Premier Clinical Research, Spokane, Washington
- Georgia (3):
  - Site 9911, Tbilisi
  - Site 9913, Tbilisi
  - Site 9912, Tbilisi
- Ukraine (7):
  - Site 3802, Dnipro
  - Site 3804, Kharkiv
  - 3808, Kharkiv
  - Site 3801, Kyiv
  - 3807, Lviv
  - Site 3803, Ternopil
  - Site 3809, Zaporizhzhya

REFERENCES:
- [Derived] Hebert A, Eichenfield L, Thiboutot D, Stein Gold L, Vassileva S, Mihaylova Y, Cartwright M, Moro L, Fragasso E, Han J, Squittieri N, Mazzetti A. Efficacy and Safety of 1% Clascoterone Cream in Patients Aged > 12 Years With Acne Vulgaris. J Drugs Dermatol. 2023 Feb 1;22(2):174-181. doi: 10.36849/JDD.7000. PMID 36745367
- [Derived] Piszczatoski CR, Powell J. Topical Clascoterone: The First Novel Agent for Acne Vulgaris in 40 Years. Clin Ther. 2021 Oct;43(10):1638-1644. doi: 10.1016/j.clinthera.2021.08.007. Epub 2021 Oct 2. PMID 34607697
- [Derived] Hebert A, Thiboutot D, Stein Gold L, Cartwright M, Gerloni M, Fragasso E, Mazzetti A. Efficacy and Safety of Topical Clascoterone Cream, 1%, for Treatment in Patients With Facial Acne: Two Phase 3 Randomized Clinical Trials. JAMA Dermatol. 2020 Jun 1;156(6):621-630. doi: 10.1001/jamadermatol.2020.0465. PMID 32320027

RESULTS

PARTICIPANT FLOW:
Groups:
- CB-03-01 Cream: CB-03-01 cream, 1% applied twice daily for 12 weeks
  Cortexolone 17α-propionate (USAN/INN: clascoterone) is a steroidal antiandrogen that is being developed as a 1% cream for the topical treatment of acne vulgaris.
Period: Overall Study
Arm/Group | CB-03-01 Cream | Vehicle Cream
Started | 353 | 355
Completed | 287 | 290
Not Completed | 66 | 65
Not completed — Lost to Follow-up | 39 | 32
Not completed — Withdrawal by Subject | 21 | 15
Not completed — Adverse Event | 3 | 6
Not completed — Withdrawal by parent | 2 | 3
Not completed — Lack of Efficacy | 0 | 3
Not completed — Noncompliance with study drug | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Progressive disease | 1 | 0
Not completed — Multiple reasons | 0 | 2

BASELINE CHARACTERISTICS:
Population: Number of participants is based on the Intent to treat dataset.
Groups:
- Total: Total of all reporting groups
Arm/Group | CB-03-01 Cream | Vehicle Cream | Total
Number analyzed (Participants) | 353 | 355 | 708
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.0 (6.7) | 19.9 (6.8) | 19.9 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221 | 215 | 436
  Male | 132 | 140 | 272
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 94 | 80 | 174
  Not Hispanic or Latino | 259 | 275 | 534
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 9 | 10 | 19
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 31 | 38 | 69
  White | 298 | 297 | 595
  More than one race | 9 | 7 | 16
  Unknown or Not Reported | 4 | 2 | 6
Baseline IGA [Count of Participants; unit: Participants] — Investigator's Global Assessment (IGA)
  Participants
    0 - Clear | 0 | 0 | 0
    1 - Almost Clear | 0 | 0 | 0
    2- Mild | 0 | 0 | 0
    3 - Moderate | 292 | 291 | 583
    4 - Severe | 61 | 64 | 125
Baseline Acne Lesion Counts [Mean (Standard Deviation); unit: Lesions]
  Non-inflammatory lesions | 59.1 (22.2) | 60.7 (22.1) | 59.9 (22.1)
  Inflammatory lesions | 42.4 (11.8) | 42.9 (12.3) | 42.7 (12.1)
  Total Lesion Count | 101.5 (25.1) | 103.6 (26.1) | 102.6 (25.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Success in Investigator's Global Assessment (IGA)
Description: Percentage of subjects in each treatment group achieving "success" at Week 12, with "success" defined as an IGA score of "clear (score=0)" or "almost clear (score=1)" and at least a two-point reduction in IGA compared to Baseline.
Time Frame: Week 12
Population: Intent-to-treat (ITT) population included all randomized subjects.
Measure: Number; unit: Percentage of participants
Arm/Group | CB-03-01 Cream | Vehicle Cream
Number analyzed (Participants) | 353 | 355
Percentage of participants | 18.4 | 9.0

2. Primary Outcome: Change From Baseline in Non-inflammatory Lesion Counts
Description: Absolute change from Baseline in non-inflammatory lesion counts in each treatment group at Week 12.
Time Frame: Baseline and Week 12
Population: ITT population.
Measure: Mean (95% Confidence Interval); unit: Non-inflammatory Lesions
Arm/Group | CB-03-01 Cream | Vehicle Cream
Number analyzed (Participants) | 353 | 355
Non-inflammatory Lesions | -19.4 [-22.6 to -16.7] | -13.0 [-15.7 to -10.3]

3. Primary Outcome: Change From Baseline in Inflammatory Lesion Counts
Description: Absolute change from Baseline in inflammatory lesion counts in each treatment group at Week 12.
Time Frame: Baseline and Week 12
Population: ITT population.
Measure: Mean (95% Confidence Interval); unit: Inflammatory Lesions
Arm/Group | CB-03-01 Cream | Vehicle Cream
Number analyzed (Participants) | 353 | 355
Inflammatory Lesions | -19.3 [-21.1 to -17.5] | -15.5 [-17.3 to -13.6]

4. Secondary Outcome: Change From Baseline in Total Lesion Counts
Description: Absolute change from Baseline in total lesions counts in each treatment group at Week 12.
Time Frame: Baseline and Week 12
Population: ITT population
Measure: Mean (95% Confidence Interval); unit: Total lesions
Arm/Group | CB-03-01 Cream | Vehicle Cream
Number analyzed (Participants) | 353 | 355
Total lesions | -39.1 [-43.0 to -35.1] | -28.8 [-32.6 to -24.9]

5. Secondary Outcome: Percent Change From Baseline in Total Lesion Counts
Description: Percent change from Baseline in total lesions counts in each treatment group at Week 12.
Time Frame: Baseline and Week 12
Population: ITT population
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | CB-03-01 Cream | Vehicle Cream
Number analyzed (Participants) | 353 | 355
percent change | -37.0 [-40.9 to -33.2] | -28.4 [-32.3 to -24.6]

6. Secondary Outcome: Percent Change From Baseline in Non-inflammatory Lesion (NIL) Counts
Description: Percent change from Baseline in non-inflammatory lesions count in each treatment group at Week 12.
Time Frame: Baseline and Week 12
Population: ITT population.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | CB-03-01 Cream | Vehicle Cream
Number analyzed (Participants) | 353 | 355
percent change | -30.6 [-35.6 to -25.7] | -21.6 [-26.4 to -16.8]

7. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion (IL) Counts
Description: Percent change from Baseline in inflammatory lesions count in each treatment group at Week 12.
Time Frame: Baseline and Week 12
Population: ITT population.
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | CB-03-01 Cream | Vehicle Cream
Number analyzed (Participants) | 353 | 355
percent change | -44.8 [-49.0 to -40.5] | -36.5 [-40.8 to -32.2]

8. Other Pre Specified Outcome: Local Site Reactions
Description: Local Site Reactions (LSRs) including telangiectasia, skin atrophy, striae rubrae, erythema, edema, scaling/dryness, stinging/burning, and pruritus scored by frequency and severity at every visit (Baseline, Weeks 4, 8, and 12).
Time Frame: Baseline, Weeks 4, 8, and 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from screening visit, Baseline (Day 1) and up to Week 12/early termination.
Description: The Safety population was used for all analyses which comprised of all participants enrolled in the study and applied at least on dose of the test article.
Arm/Group | CB-03-01 Cream | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/353 | 0/355
Serious Adverse Events (participants affected / at risk) | 0/353 | 1/355
Other Adverse Events (participants affected / at risk) | 9/353 | 18/355
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CB-03-01 Cream (N=353) | Vehicle Cream (N=355)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — The SAE was deemed not related to test article.
OTHER ADVERSE EVENTS (reported when occurring in more than 0.6% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CB-03-01 Cream (N=353) | Vehicle Cream (N=355)
Nasopharyngitis (Infections and infestations) | 6 (7) | 12 (12)
Application pain (General disorders) | 1 (1) | 3 (4)
Application site pruritus (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to publish pooled study data. In the event that such manuscript has not been submitted for publication within 18 months from study completion/termination at all participating sites, the PI shall have the right to single center publications provided they submit any data for presentation, oral or written, to the Sponsor for review 60 days prior to public disclosure. The PI may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-08-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT02608450/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT02608450/SAP_001.pdf